CLINICAL TRIAL: NCT01594294
Title: EVALUATION OF THE EFFECTS OF CLEAR CARE® / AOSEPT® PLUS HYDROGEN PEROXIDE SOLUTION ON THE EYELID TISSUES - Part III: COMPARATIVE EVALUATION WITH RENU® MPS OVER 3 MONTH OF WEAR - CONTROL EVALUATION WITH AIR OPTIX® AQUA and ACUVUE® 2®
Brief Title: An Evaluation of Marketed Contact Lens Disinfectant Systems on Eyelid Tissues
Acronym: ID11-56
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alcon Research (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: M-11-09
Record Dates: First submitted 2012-05-07; First posted 2012-05-09 (Estimated); Results first posted 2014-07-25 (Estimated); Last update posted 2014-07-25 (Estimated); Status verified 2014-06

CONDITIONS: Myopia
Keywords: CLEAR CARE®; AOSEPT® Plus; ReNu MultiPlus®; silicone hydrogel; hydrogel; ACUVUE® 2®; AIR OPTIX® AQUA; eyelid response; wettability; contamination; contact lenses
MeSH Terms: conditions — Myopia

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- AOSEPT Plus (Experimental): AOSEPT® Plus contact lens solution used with etafilcon A contact lenses or lotrafilcon B contact lenses for 3 months (Investigational Phase)
  Interventions: Device: AOSEPT® Plus contact lens solution; Device: Etafilcon A contact lenses; Device: Lotrafilcon B contact lenses
- ReNu MultiPlus (Active Comparator): ReNu MultiPlus® contact lens solution used with etafilcon A contact lenses or lotrafilcon B contact lenses for 3 months (Investigational Phase)
  Interventions: Device: ReNu MultiPlus® contact lens solution; Device: Etafilcon A contact lenses; Device: Lotrafilcon B contact lenses
- Complete MPS Easy Rub (Other): COMPLETE® MPS Easy Rub® Formula contact lens solution used with etafilcon A contact lenses (14 days) or lotrafilcon B contact lenses (30 days), Screening Phase
  Interventions: Device: Etafilcon A contact lenses; Device: Lotrafilcon B contact lenses; Device: COMPLETE® MPS Easy Rub® Formula contact lens solution

INTERVENTIONS:
Device: AOSEPT® Plus contact lens solution — Hydrogen peroxide-based cleaning and disinfection system
  Other Names: CLEAR CARE®
  Arms: AOSEPT Plus
Device: ReNu MultiPlus® contact lens solution — Polyaminopropyl biguanide (PHMB) preserved multipurpose solution
  Arms: ReNu MultiPlus
Device: Etafilcon A contact lenses — Hydrogel contact lenses worn on a daily wear basis for 14 days (Screening Phase) and 3 months (Investigational Phase). During the Investigational Phase, the contact lenses lenses were worn a minimum of six hours per day, 5 days per week, with a fresh pair dispensed every 2 weeks.
  Other Names: ACUVUE® 2®
Device: Lotrafilcon B contact lenses — Silicone hydrogel contact lenses worn on a daily wear basis for 30 days (Screening Phase) and 3 months (Investigational Phase). During the Investigational Phase, the contact lenses lenses were worn a minimum of six hours per day, 5 days per week, with a fresh pair dispensed monthly.
  Other Names: AIR OPTIX® AQUA
Device: COMPLETE® MPS Easy Rub® Formula contact lens solution — PHMB 0.0001% and poloxamer 0.05% multipurpose solution
  Arms: Complete MPS Easy Rub

SUMMARY:
The purpose of this study was to assess and compare the effect of the repeated usage of 2 different care systems (one hydrogen peroxide based cleaning and disinfecting system and one PHMB containing multipurpose system) with ACUVUE® 2® and AIR OPTIX® AQUA contact lenses worn on a daily wear basis for a 3-month period.

DETAILED DESCRIPTION:
This study was divided into 2 periods, a Screening Phase and an Investigational Phase. During the Screening Phase, subjects were fitted and dispensed with either ACUVUE® 2® (for current hydrogel wearers) or AIR OPTIX® AQUA (for current silicone hydrogel wearers) contact lenses and used COMPLETE® MPS Easy Rub® Formula to clean and disinfect their lenses. At the completion of the Screening Phase, the symptomatic status of the subjects was re-assessed. Those subjects who qualified proceeded to the Investigational Phase and were dispensed with new pair of study contact lenses identical to the lenses they wore during the Screening Phase to use in conjunction with the allocated study care product, CLEAR CARE® /AOSEPT® Plus or ReNu MultiPlus®.

ELIGIBILITY:
Inclusion Criteria:

* Read and understand the Participant Information Sheet;
* Read, sign, and date an Informed Consent;
* Successfully wearing a frequent replacement hydrogel or silicone hydrogel contact lens brand under a frequent replacement (biweekly or monthly) daily wear modality;
* Classified as symptomatic according to protocol-specified criteria;
* Agree to wear study contact lenses as directed for the duration of the study;
* Best corrected visual acuity (BCVA) of 6/9 or better in each eye;
* Other protocol-defined inclusion criteria may apply.

Exclusion Criteria:

* Any known sensitivity or intolerance to any of the contact lenses or contact lens care products to be used;
* Monocular vision (only one eye with functional vision or only one eye fitted with contact lenses);
* History of seasonal allergies, which may have an adverse impact on contact lens wear, or data and information obtained in this study;
* Systemic disease or use of medication which might interfere with contact lens wear or produce dry eye side effects;
* Ocular allergies or ocular disease which might interfere with contact lens wear or data and information obtained in this study;
* Active ocular infection;
* Use of any concomitant topical ocular medications during the study period;
* Significant ocular anomaly;
* Previous ocular surgery;
* History of recent, significant changes in visual acuity;
* Any medical condition that might be prejudicial to the study;
* Pregnant, planning to be become pregnant, or lactating at time of enrollment;
* Any infectious disease (e.g. hepatitis, tuberculosis), immunosuppressive disease (e.g. HIV), or diabetes;
* Participation in an investigational drug or device study within 30 days of entering study;
* Other protocol-defined exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2012-04; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Renee Garofalo, OD, FAAO, Study Director — Alcon Research

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Of the 100 participants enrolled, 21 were exited as screen failures prior to initiation of the Investigational Phase. This reporting group includes all participants randomized into the Investigational Phase (79).
Period: Overall Study
Arm/Group | AOSEPT Plus | ReNu MultiPlus
Started | 39 | 40
Completed | 36 | 36
Not Completed | 3 | 4

BASELINE CHARACTERISTICS:
Population: This analysis population includes all participants who completed the study as per the protocol.
Groups:
- Total: Total of all reporting groups
Arm/Group | AOSEPT Plus | ReNu MultiPlus | Total
Number analyzed (Participants) | 35 | 36 | 71
Age, Continuous [Mean (Standard Deviation); unit: years] | 35.7 (11.1) | 37.1 (10.7) | 36.4 (10.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21 | 25 | 46
  Male | 14 | 11 | 25

OUTCOME MEASURES:

1. Primary Outcome: Maximum Papillae
Description: Eyelid papillae (bumps on the inner eyelid) were recorded separately for three zones of the upper lid and overall for the lower lid on a 5-point forced choice scale: 0 = None; 1 = Slight (diffuse papillae); 2 = Mild (diffuse & tufts papillae); 3 = Moderate (moderate & tufts papillae); 4 = Severe (giant papillae). The maximum value represents the worse grade in any zone. Both eyes were included in the model for analysis. Contact lenses were not worn for this assessment.
Time Frame: Baseline (Day 0), Month 3
Population: This analysis population includes all participants who completed the study as per the protocol, minus missing responses.
Measure: Median (Full Range); unit: Units on a scale
Units Other Than Participants: Eyes
Arm/Group | AOSEPT Plus | ReNu MultiPlus
Number analyzed (Participants) | 35 | 36
Number analyzed (Eyes) | 68 | 71
Units on a scale
  Baseline (Day 0) | 1.50 [.50 to 3.00] | 1.00 [.00 to 3.00]
  Month 3 | 1.50 [.50 to 3.00] | 1.00 [.00 to 3.00]

2. Primary Outcome: Maximum Eyelid Hyperaemia
Description: Eyelid hyperaemia (redness) was recorded separately for three zones of the upper lid and overall for the lower lid on a 5-point forced choice scale: 0 = Clear; 1 = Slight redness; 2 = Mild redness; 3 = Moderate redness; 4 = Severe redness). The maximum value represents the worst grade in any zone. Both eyes were included in the model for analysis. Contact lenses were not worn for this assessment.
Time Frame: Baseline (Day 0), Month 3
Population: This analysis population includes all participants who completed the study as per the protocol, minus missing responses.
Measure: Median (Full Range); unit: units on a scale
Units Other Than Participants: Eyes
Arm/Group | AOSEPT Plus | ReNu MultiPlus
Number analyzed (Participants) | 35 | 36
Number analyzed (Eyes) | 68 | 71
units on a scale
  Baseline (Day 0) | 2.00 [1.00 to 3.00] | 2.00 [1.00 to 3.50]
  Month 3 | 2.00 [1.50 to 4.00] | 2.00 [1.00 to 3.00]

3. Primary Outcome: Mean Upper Eyelid Redness
Description: The contact lenses were removed and upper eyelid redness was objectively measured through digital images. The coverage of the palpebral surface by blood vessels is expressed as percentage of the total surface measured. Both eyes were included in the model for analysis. Contact lenses were not worn for this assessment.
Time Frame: Baseline (Day 0), Month 3
Population: This analysis population includes all participants who completed the study as per the protocol, minus missing responses.
Measure: Mean (Standard Deviation); unit: percentage of total surface measured
Units Other Than Participants: Eyes
Arm/Group | AOSEPT Plus | ReNu MultiPlus
Number analyzed (Participants) | 35 | 36
Number analyzed (Eyes) | 68 | 71
percentage of total surface measured
  Baseline (Day 0) | 34.7 (15.5) | 31.9 (9.1)
  Month 3 | 33.4 (13.4) | 30.8 (12.7)

4. Primary Outcome: Mean Upper Eyelid Margin Staining
Description: The contact lens was removed and ophthalmic dye was instilled. Upper eyelid margin staining was objectively measured through digital images. The extent of true staining (i.e., the total area of lid margin covered by staining) was recorded. Both eyes were included in the model for analysis. Contact lenses were not worn for this assessment.
Time Frame: Baseline (Day 0), Month 3
Population: This analysis population includes all participants who completed the study as per the protocol, minus missing responses.
Measure: Mean (Standard Deviation); unit: square millimeters
Units Other Than Participants: Eyes
Arm/Group | AOSEPT Plus | ReNu MultiPlus
Number analyzed (Participants) | 35 | 36
Number analyzed (Eyes) | 68 | 71
square millimeters
  Baseline (Day 0) | 5.36 (4.21) | 4.33 (2.65)
  Month 3 | 4.49 (2.90) | 4.80 (2.82)

5. Secondary Outcome: Median Non-Invasive Pre-Lens Tear Film Break Up Time (PL-NIBUT)
Description: The pre-lens tear film is the layer of tears located on top of the contact lens (i.e., between the eyelid and the contact lens). The time required for a dry spot to appear on the pre-lens surface after blinking is referred to as the pre-lens tear film break up time. PL-NIBUT was evaluated using a biomicroscope with a diffuse illumination source, i.e., Tearscope. A longer PL-NIBUT indicates a more stable tear film and greater on-eye lens wettability. Three PL-NIBUT measurements were recorded, and the median value was used for analysis. Both eyes were included in the model for analysis. Contact lenses were on-eye for this assessment.
Time Frame: Month 3
Population: This analysis population includes all participants who completed the study as per the protocol, minus missing responses.
Measure: Mean (Standard Deviation); unit: seconds
Units Other Than Participants: Eyes
Arm/Group | AOSEPT Plus | ReNu MultiPlus
Number analyzed (Participants) | 35 | 36
Number analyzed (Eyes) | 68 | 71
seconds | 4.16 (3.50) | 4.52 (3.46)

ADVERSE EVENTS:
Time Frame: Adverse events were collected for the duration of the study (April 2012 to June 2013). An adverse event was any untoward medical occurrence in a subject administered a test article regardless of causal relationship with the treatment.
Description: This analysis population includes all participants exposed to the test product during the Investigational Phase.
Arm/Group | AOSEPT Plus | ReNu MultiPlus
Serious Adverse Events (participants affected / at risk) | 2/39 | 2/39
Other Adverse Events (participants affected / at risk) | 3/39 | 0/39
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | AOSEPT Plus (N=39) | ReNu MultiPlus (N=39)
Fall causing crack on the skull and internal bleeding (Injury, poisoning and procedural complications) | 1 | 0
Fibroids (Surgical and medical procedures) | 1 | 0
Hernia (Surgical and medical procedures) | 0 | 1
Dehydration and possible chest infection (Surgical and medical procedures) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | AOSEPT Plus (N=39) | ReNu MultiPlus (N=39)
Toxic reaction (Injury, poisoning and procedural complications) | 3 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor reserves the right of prior review of any publication or presentation of information related to the study.